CLINICAL TRIAL: NCT00208429
Title: Uncontrolled Prospective Multi-Centre Post Marketing Surveillance Study to Monitor the Long Term Survivorship of Pinnacle Acetabular Cup System With a Metal on Enduron Polyethylene Bearing in Subjects With Aetiologies Requiring a Primary Total Hip Replacement
Brief Title: A Multi-centre Study to Assess the Long-term Performance of the Pinnacle™ Cup With a Polyethylene-on-metal Bearing in Primary Total Hip Replacement
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Site Principal Investigator became seriously ill, so study abandoned before the start of recruitment
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT03/40
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Post-traumatic Arthritis; Collagen Disorders; Avascular Necrosis; Traumatic Femoral Fractures; Nonunion of Femoral Fractures; Congenital Hip Dysplasia; Slipped Capital Femoral Epiphysis
Keywords: Hip; Cementless
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Collagen Diseases; Osteonecrosis; Hip Dislocation, Congenital; Slipped Capital Femoral Epiphyses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pinnacle Acetabular System (Other)
  Interventions: Device: Pinnacle Acetabular System

INTERVENTIONS:
Device: Pinnacle Acetabular System

SUMMARY:
The purpose of this study is to monitor the performance of the Pinnacle™ Cup with a polyethylene-on-metal bearing combination in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be evaluated at regular intervals following hip surgery using patient, clinical and x-ray assessments.

ELIGIBILITY:
Inclusion Criteria:

i) Male or female subjects, aged between 18 and 70 years inclusive.

ii) Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.

iii) Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

iv) Subjects undergoing primary total hip replacement who are suitable for a cementless acetabular component and a metal on polyethylene bearing.

Exclusion Criteria:

i) Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.

ii) Subjects undergoing revision hip replacement.

iii) Subjects undergoing simultaneous bilateral hip operation.

iv) Subjects with a contralateral hip replacement, which was implanted less than six months previously or is not performing satisfactorily.

v) Women who are pregnant.

vi) Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.

vii) Subjects who have participated in a clinical study with an investigational product in the last 12 months.

viii) Subjects who are currently involved in any injury litigation claims.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-07-01 (Actual); Primary Completion 2009-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Kaplan-Meier survivorship calculated at the five-year time-point. | 5 yrs post surgery

SECONDARY OUTCOMES:
Change in Baseline to post-operative assessment in clinical outcome using the Harris Hip Score | 6mths, 1yr, 2yrs, 5yrs, 7yrs, 10yrs and 15yrs post-surgery
Change in Baseline to post-operative assessment in clinical outcome using the Oxford Hip Score | Annually up to 15 yrs post-surgery
Kaplan-Meier survivorship | Annually up to 15 yrs post-surgery